CLINICAL TRIAL: NCT07038694
Title: A New Rehabilitation Language: Understanding Adoption of the Rehabilitation Treatment Specification System Into Physiotherapists Documentation
Brief Title: RTSS Adoption Into Physiotherapists Documentation
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 12584
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Rehabilitation; Clinical Reasoning; Medical Record Documenation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rehabilitation physiotherapy RTSS users: Physiotherapists will be recruited exclusively from the rehabilitation department of physiotherapy at Guy's and St Thomas' hospital,. Purposive, maximum variation sampling will be used to sample physiotherapists who have attempted adoption of RTSS into clinical notes. Applying Malterud et al's concept of information power suggests an estimated sample of 12-16 participants will be required, calculated from the study's narrow aim, the specificity of the sample with respect to the aim, the application of theory and encouragement of strong dialogue via an interviewer experienced in the subject. Purposive maximum variation sampling will ensure heterogeneity of clinical experience (Agenda for Change (AFC) bandings 3-8) to support diversity of perspectives and experiences for data analysis.
  Interventions: Other: Qualitative semi structured interview

INTERVENTIONS:
Other: Qualitative semi structured interview — 60 minute, virtually performed via Microsoft Teams, semi-structured interview

SUMMARY:
The Rehabilitation Treatment Specification System (RTSS) is a framework that aims to support clinicians in reasoning and documenting how to deliver rehabilitation. This was explored in a pilot study in 2023 that tested the feasibility of a 6-week teaching programme aiming to support the adoption of the RTSS into practise of physiotherapists and subsequently measure its effect on clinicians reasoning of treatment. Whilst clinical reasoning scores improved, adoption of the framework remained low. Interviews within this study revealed the difficulty clinicians experienced in transitioning to documenting the RTSS.

Further local work within Guy's & St Thomas NHS foundation trust (GSTT) resulted in modified integrations of the RTSS into electronic health record systems as well as training, yet adoption still remained limited. With documentation being cited as an influence of RTSS adoption and thus contributing to its clinical benefit, this qualitative study will attempt to make clear what factors facilitate and/or limit RTSS documentation adoption, and how they exert their influence. The findings from this study will inform the design of interventions that will aid future study of benefit of the RTSS on physiotherapy practice.

To achieve these aims, interviews will be conducted virtually via MS Teams, by the lead researcher, with approximately 12-16 volunteering physiotherapists who have attempted to document the RTSS, within the site of GSTT. The interviews will last approximately 1 hour, and will be partially structured in nature to invite in-depth discussion of topic. Analyses of the data will be performed by a team of 3 clinical academics working between GSTT and King's College London with study findings to be disseminated in a peer-reviewed journal and at professional conferences

DETAILED DESCRIPTION:
Rehabilitation frameworks, such as the international classification of functioning, disability and health, 1 support the reasoning and identification of what should be targeted by clinicians to achieve desired patient outcomes. However, frameworks supporting the reasoning about how these targets should be treated are scarce. A promising candidate that provides this function is the rehabilitation treatment specification system (RTSS) 2. The RTSS encourages clinicians to hypothesise a claim (a treatment theory) about how they are going to treat an individual patient by identifying treatment components - the tripartite building block of a specified treatment composed of a singular (measurable) treatment target i.e., an aspect of function or disability that is to be changed directly by the ingredient(s), 1 or more (measurable) ingredients i.e., what the clinician does to modify the target, and the mechanism(s) of action (MoA) i.e., the causal chain through which the treatment is known or hypothesised to work (i.e. how the ingredients affect the target) 3. Proponents of the RTSS hypothesised that by facilitating clinicians to explicate their treatment theory, their treatment reasoning would develop 4. We explored this hypothesis in a first-phase pilot study which assessed whether a 6-week multi-modal RTSS teaching programme was feasible and had any effect on a small group of clinicians' clinical reasoning 5. We observed an improvement in self-reported measures of clinical reasoning despite the targeted behaviour (clinical uptake of the RTSS) remaining low. Critically, nested qualitative data revealed the difficulty clinicians experienced in transitioning to documenting the RTSS, citing the need for documenting training and more integrative electronic medical record (EMR) systems. Since the publication of this work, a quality improvement project within Guy's & St Thomas' NHS foundation trust has seen the design and implementation of an RTSS EMR integration which physiotherapists have attempted to adopt.

Clinicians concur with the concept that documentation practices can enhance clinical reasoning and quality of care 6. They also report documenting as becoming increasingly burdensome, with a need to satisfy evolving legislative, funding and medico-legal purposes 7, 8 resulting in clinicians' time spent documenting becoming similar to time spent providing clinical care 9. As well as navigating the multitude of purposes, clinicians cite a number of personal and environmental factors that contribute to their documenting practices 10. If not considered, these can lead to non-adoption. For example one study concluded that a novel documenting practice for physiotherapists was infeasible due to time requirements, differing personal and interpersonal cultures, disagreements with the EMR structure, and a lack of organisational support and motivation 11. Thus, contextual exploration of the lived experience of physiotherapists attempting to adopt an RTSS EMR integration is imperative to better understand adoption behaviours and inform development of strategies that could enhance adoption.

This is a student project as part of a Masters in Clinical Research (MRes) course. Through critically exploring the experience of clinical physiotherapists attempting to adopt RTSS documentation practices through a framework analysis method, valuable insight will be provided on what and how determinants modulate RTSS documentation adoption, and inform implementation interventions that seek to utilise the RTSS in physiotherapy, and rehabilitation practice.

* The aim of this study is to explore attitudes and perceptions regarding the implementation of the RTSS into documentation practises of physiotherapists working in a hospital setting
* The primary objectives of this study are:

  * To explore perceived facilitators to adoption of the RTSS into physiotherapists documentation practice
  * To explore perceived barriers to adoption of the RTSS into physiotherapists documentation practices
  * To understand how facilitators and barriers exert their influence on physiotherapists behaviours of adopting the RTSS into their documentation practices
  * To identify implementation interventions that may support the behaviour of adopting the RTSS into documentation practices

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapy staff who have attempted adoption of the RTSS documentation integration
* Are actively working in the physiotherapy department setting with in substantive positions

Exclusion Criteria:

* Are unable to consent to the study
* Are student physiotherapists or temporary staff
* Are actively working with the PI
* Are unable to conduct the interview in English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physiotherapists will be recruited exclusively from the rehabilitation department of physiotherapy at Guy's and St Thomas' hospital, these are physiotherapists who have attempted to use the RTSS in clinical documentation.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Semi Structured qualitative Interview | From early July 2025 to end of July 2025
  Semi structured qualitative interviews performed via MS Teams lasting up to 1 hour in duration

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hart T, Dijkers MP, Whyte J, Turkstra LS, Zanca JM, Packel A, Van Stan JH, Ferraro M, Chen C. A Theory-Driven System for the Specification of Rehabilitation Treatments. Arch Phys Med Rehabil. 2019 Jan;100(1):172-180. doi: 10.1016/j.apmr.2018.09.109. Epub 2018 Sep 27. PMID 30267669